CLINICAL TRIAL: NCT05909800
Title: Randomized, Double-blind, Multicenter, Parallel-group, Placebo-controlled Study to Evaluate the Efficacy of Phenofibrate Treatment on the Functions of Beta Cells in Children and Adolescents With Newly Diagnosed of Type 1 Diabetes.
Brief Title: Prolonged Remission Induced by Phenofibrate in Children Newly Diagnosed With Type 1 Diabetes.
Acronym: PRIFEN
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Collaborators: Children's Memorial Health Institute, Poland (Other)
Responsible Party: Principal Investigator, AGNIESZKA SZYPOWSKA, Deputy Head of the Clinical Department of Pediatric Diabetology and Pediatrics, Medical University of Warsaw
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRIFEN-01; 2020-003916-28 (EudraCT Number)
Record Dates: First submitted 2022-11-29; First posted 2023-06-18 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes Mellitus; sulfatide; phenofibrate; children; adolescents; randomized controlled trial; fenofibrate
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — Fenofibrate

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to two groups, receiving either phenofibrate at a dose of 160 mg or placebo, orally, once daily, for 12 months. All study participants will be followed up for up to 12 months after the start of the intervention. Study visits at month 3, 6, 9 and 12 will be coordinated with diabetes outpatient clinic visits.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, caregivers, investigators, outcome assessors, and the person responsible for the statistical analysis will be blinded to the intervention until completion of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phenofibrate (Experimental): Phenofibrate in capsules received orally, daily, for 12 months.
  Interventions: Drug: Phenofibrate
- Placebo (Placebo Comparator): Capsules containing Microcrystalline cellulose 102,594 mg (99%) and Magnesium stearate 6 mg (1%) identical to those of the active product received orally, daily, for 12 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Phenofibrate — Administred orally, once daily, for 12 months.
  Other Names: Fenofibrate; Fenofibratum; SUB07576MIG; CAS no. 49562-28-9
  Arms: Phenofibrate
Drug: Placebo — Administred orally, once daily, for 12 months.
  Other Names: inactive drug; inactive medicine; inactive substance.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to evaluate of the effect of phenofibrate on the functions of beta cells in children with new diagnosis of type 1 diabetes. The main question it aims to answer is: whether phenofibrate may prolong residual beta-cell function therefore own insulin secretion. Participants will be asked to take a phenofibrate or identically appearing placebo (a neutral substance), orally, once daily, for 12 months with no knowledge what is administred to them. They will be invited for follow-up visits including blood tests every 3 months. Researchers will be monitoring the two groups for the safety of the phenofibrate, and at the trial end they compare the residual insulin secretion results in two groups.

DETAILED DESCRIPTION:
Rationale:

Preservation of residual pancreatic beta cell function in children with newly diagnosed T1D gives a chance for better diabetes control, reduction of chronic diabetes complications, and possibly temporary insulin withdrawal. Indication of a cheap drug for secondary prevention of T1D.

Setting:

Recruitment will be through the paediatric diabetes clinics at two participating centres in Warsaw, Poland (Department of Paediatrics, the Medical University of Warsaw and Department of Endocrinology and Diabetology, Children's Memorial Health Institute).

The initiation of study treatment may be performed no later than 28 days after screening visit, and no later than in 8 weeks from diabetes diagnosis.

PICO:

Adolescent participants meeting inclusion criteria, newly diagnosed with type 1 diabetes will be randomly assigned to two groups, receiving either fenofibrate at a dose of 160 mg or placebo, and regularly assesed, every 3 months for the next year. Assuming increase by 50% of AUC of C-peptide in the test group compared to placebo, 88 subjects are needed to achieve power of 85%. If about 13% drop-out is assumed the total group size is 102 patients. Given randomization ratio 1:1, there is 51 patients in each group.

Main study procedures:

* Demographic and medical history.
* Physical examination and vital signs: heart rate and blood pressure, respiration rate, body temperature.
* Blood collection for laboratory analysis (hematology: morphology with automatic blood smear, biochemistry: ALT, AST, total bilirubin, albumin, amylase, lipase, total cholesterol, HDL, LDL, triglycerides, GGTP, HbA1c, TSH, FT4, Anti-Tg, Anti-TPO, CK, creatinine, urea, vitamin D, homocysteine, Anti-tTG IgA, IgA.
* Urine pregnancy test (in girls with childbearing potential).
* C-peptide and Glucose in MMTT stimulation assay.
* Anti-insulin IAA antibodies, Antibodies to glutamic acid decarboxylase (GADA), Antibodies to tyrosine phosphatase (IA2A), Antibodies to the zinc transporter 8 (ZnT8).
* IL1, IL2, IL10.
* TNF alpha, IFN gamma.
* Genetic study - WES genome sequencing, HLA DR3, DR4, DO8, DQ7.
* FGM Libre Free Style Glucose Monitoring System.
* Abdominal ultrasound.
* Ultrasound of the thyroid gland.
* Safety monitoring and AE collection.
* IMP administration. Compliance will be assessed by collecting empty packages as well as by direct interview and participants receiving <75% of the recommended doses will be considered as non-compliant.

ELIGIBILITY:
Inclusion Criteria:

Subjects who meet all of the following criteria are eligible to participate in this study:

1. Subject or Legally accepted representative (LAR) able to understand and provide signed informed consent. Assent is also required of adolescents and children.

   * LAR of subjects ≤ 17 years sign the "Information Leaflet and ICF for the Parent/Legal Guardian of Minor Subject".
   * Adolescents from 10-15 years sign "Children Assent form".
   * Adolescents from 16-17 years sign "Adolescent Assent form".
2. Age ≥10 and ≤ 17 years.
3. Diagnosis of type 1 diabetes within 8 weeks before randomization (V0 visit) based on positive autoantibody (minimum 1 among: GADA, IA2A, ZnT4, IAA) and symptoms of type 1 diabetes according to the criteria of the Polish Diabetes Association (1 of the following):

   * symptoms of diabetes and blood glucose ≥ 200 mg / dl (≥ 11.1 mmol/l),
   * when no symptoms or when diabetes symptoms are present and random glucose <200 mg/dl (<11.1 mmol/l) - then confirmation of the diagnosis is fasting blood glucose in 2 measurements ≥ 126 mg/dl (≥ 7.0 mmol/l); each test must be performed on a different day,
   * in the absence of symptoms of hyperglycaemia and random glycaemia ≥ 200 mg/dl (11.1 mmol/l), fasting glucose ≥ 126 mg/dl (7.0 mmol/l) is a confirmation of the diagnosis,
   * if once or twice fasting blood glucose is 100-125 mg / dl (5.6-6.9 mmol/l), or if fasting blood glucose is below 100 mg/dl (5.6 mmol/l) ) exists, If there is a reasonable suspicion of impaired glucose tolerance or diabetes mellitus, an oral glucose tolerance test (OGTT) should be performed. At the 120th minute of the OGTT, blood glucose ≥ 200 mg/dl (11.1 mmol/l) confirms the diagnosis of diabetes.
4. Male or nonpregnant and nonlactating female who is abstinent or agrees to use effective contraceptive methods throughout the course of the study. Acceptable birth control methods are the following:

   * Intrauterine device in place for at least 3 months.
   * Use of condom or diaphragm with spermicide for at least 14 days prior to the Visit 0 visit and through study completion.
   * Stable hormonal contraceptive for at least 2 months prior to the Visit 0 and continuing through study completion.
5. Females (menstruating) must have a negative urine beta-human chorionic gonadotropin hormone (hCG) pregnancy test at Visit 0.

Exclusion Criteria:

Subjects who meet any of the following criteria are not eligible to participate in this study:

1. Age under 10 or over 17.
2. Lack of consent of at least one the guardian LAR to participate in the study.
3. Treatment with any oral or injected anti-diabetic medications other than insulin.
4. The Subject or close Subject's family history, past or present of allergic or hypersensitivity reactions to fenofibrate or any of the excipients (including patients with hereditary problems of galactose intolerance, total lactase deficiency or glucose-galactose malabsorption).
5. Severe hypersensitivity reaction to any other drug.
6. Subjects with current or history of clinically significant renal impairment.
7. Subjects with current or history of clinically significant hepatic impairment.
8. Subjects with or history of significant gastrointestinal disease including celiac disease, gastroparesis, another disorder of intestinal absorption or motility.
9. Subject with current or history of gall bladder disease.
10. Present or history of chronic or acute pancreatitis, except acute pancreatitis due to severe hypertriglyceridaemia.
11. Photosensitivity or phototoxic reactions after the use of fibrates or chemically related substances, e.g. ketoprofen.
12. Subjects who tested positive for pregnancy at screening and V0 visit or who are currently breastfeeding.
13. Low blood albumin defined as clinically significant by investigator.
14. Patients with pre-disposing factors for myopathy and/or rhabdomyolysis, including personal and familial history of hereditary muscular disorders. Unexplained persistent elevated creatine phosphokinase levels considered clinically significant by the investigator.
15. The presence of circumstances that the Investigator considers problematic when obtaining informed consent or meeting the study guidelines, or that may invalidate the interpretation of test results or expose Subjects to unnecessary risk.
16. Inability or unwillingness to comply with study procedures.
17. Any medical condition or treatment the Investigator believes may expose the Subject to unnecessary risk during the study.
18. Participation in interventional or other drug research studies which could affect the objectives of this study.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 102 (Estimated)
Dates: Start 2022-09-29 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Differences in AUC in C-peptide stimulation test | 12 months
  Assessment of pancreatic beta cell function by comparing the area under the curve (AUC) in the C-peptide stimulation test: Change in the mean insulin secretion measured on the basis of the C-peptide area under the curve in the stimulation test

SECONDARY OUTCOMES:
Differences in C-peptide concentration in the stimulation test: change in the insulin secretion measured on the basis of the fasting C-peptide concentration | 0, 6, 12 months
  Fasting C-peptide concentration in the stimulation test
Differences in parameters of diabetes control | 0,3,6,9,12 months
  HbA1c
Daily insulin requirement | 0,3,6,9,12 months
  Daily insulin requirement/kg of body mass
Interleukins | 0,6,12 months
  IL1, IL2, IL10, TNF alpha, IFN gamma
Adverse Events occurence | 0,3,6,9,12 months
  Safety will be evaluated through assessment of AEs, vital signs, physical examinations, USG findings, and laboratory evaluations. Any clinically significant laboratory occurring after study drug initiation must be reported by the investigator as an AE and/or SAE, as appropriate, and must be followed by additional laboratory evaluations until they return to normal range, stabilize, or until the change is no longer clinically relevant. All safety analyses will be conducted using the Safety Analysis Set. Adverse event data will be presented and tabulated according to MedDRA classification.
Differences in C-peptide concentration in the stimulation test: change in the insulin secretion measured on the basis of the fasting C-peptide concentration | 0,6,12 months
  Maximum C-peptide concentration
Diabetes control and glucose fluctuations | 0,3,6,9,12 months
  Mean blood glucose with standard deviation
Differences in glucose fluctuations | 0,3,6,9,12 months
  Glucose variability index (CV%)
Parameter of glucose fluctuations | 0,3,6,9,12 months
  Time in range 70-180mg/dl
Difference in autoantibodies | 0,6,12 month
  Difference in anti-insulin IAA antibodies, antibodies against glutamic acid decarboxylase (GADA), antibodies to tyrosine phosphatase (IA2A), anti-zinc transporter antibodies 8 determination.
Genetical analysis | 1 per study
  WES Whole Exome Sequencing and HLA

CONTACTS AND LOCATIONS:
Overall Officials: Agnieszka Szypowska, MD, PhD,Prof, Principal Investigator — Medical University of Warsaw
Locations (2):
- Poland (2):
  - Clinical department of pediatric diabetology and paediatrics, DSK UCKWUM, Warsaw, Masovian Voivodeship
  - Diabetology Department, Children's Memorial Health Institute, Warsaw, Masovian Voivodeship

IPD SHARING:
Plan to Share IPD: Yes
The data relevant to the study will be included in the article or uploaded as supplementary information
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Avaliable with the publication
Access Criteria: open access - web adress will be known after the publication of the paper